CLINICAL TRIAL: NCT06986551
Title: Remineralization Potential of PRG Barrier Coat Versus Fluoride Varnish in White Spot Lesions in Permanent Anterior Teeth of Children (A Randomized Controlled Trial)
Brief Title: Remineralization Potential of PRG Barrier Coat Versus Fluoride Varnish in White Spot Lesions in Permanent Anterior Teeth of Children
Acronym: PRG Barrier
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hanaa Hamdy Mohamed Fathy Mahmoud Rady, dentist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRG Barrier Remineralization
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: White Spot Lesion of Tooth; Demineralization
Keywords: PRG Barrier Coat; white spot lesion; Fluoride Varnish
MeSH Terms: interventions — PRG Barrier Coat

STUDY DESIGN:
Intervention Model Description: A random sequence will be generated by the assistant supervisor using the online form Using four-folded numbered paper on which remineralizing agent will be written contained in the closed white envelope When a patient agrees to participate in the trial, an envelope will be drawn by co-supervisor and name, telephone number and patient's I.D. will be written on it. Those selected envelopes will be opened at the treatment visit after taking baseline clinical data to choose which material should be used. Randomization and allocation concealment will be performed by the co-supervisor to avoid selection bias
Who Masked: Participant, Outcomes Assessor
Masking Description: The blinding of the operator is not possible due to the nature of the material used. Trial participants, outcome assessors and statisticians will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRG Barrier coat (Experimental): Before the application of the varnish, teeth were cleaned using a prophylaxis polishing past with a low-speed cone brush in a contra-angle low-speed handpiece. It was then dried with air and isolated using cotton rolls According to the manufacturer's instructions, for the application of PRG barrier coat varnish, a drop of the active will be mixed with the base using the attached brush. After isolation with cotton rolls, the brush will be used to smear the WSLs with the mix. I will be undisturbed for at least three seconds, then cured for 10 seconds using the visible-light curing unit.
  And there will be no postoperative instruction to the patient after application (light-cured resin material).
  Interventions: Other: PRG Barrier coat
- 5% NaF fluoride varnish (Active Comparator): Before the application of the varnish, teeth were cleaned using a prophylaxis polishing past with a low-speed cone brush in a contra angle low-speed handpiece. It will be dried with air and isolated using cotton rolls.
  Package will be unpacked, and the application guide will be used to display the contents and mix to avoid the separation of sodium fluoride components. After isolation, a thin layer of the varnish will coat . The participants will be asked to keep their mouths closed to allow the varnish to set in the presence of saliva. Rinsing or suction was not allowed immediately after the application of the varnish.
  The participants will be asked to avoid consumption of rough and viscid food or hot drinks for two hours after application of the varnish. For the rest of that day, participants will be asked to eat soft food and stop tooth brushing (Ezzeldin et al., 2024
  Interventions: Other: 5% NaF fluoride varnish

INTERVENTIONS:
Other: 5% NaF fluoride varnish — Before the application of the varnish, teeth were cleaned using a prophylaxis polishing past with a low-speed cone brush in a contra angle low-speed handpiece. It will be dried with air and isolated using cotton rolls.
  Package will be unpacked, and the application guide will be used to display the contents and mix to avoid the separation of sodium fluoride components. After isolation, a thin layer of the varnish will coat . The participants will be asked to keep their mouths closed to allow the varnish to set in the presence of saliva. Rinsing or suction was not allowed immediately after the application of the varnish.
  The participants will be asked to avoid consumption of rough and viscid food or hot drinks for two hours after application of the varnish. For the rest of that day, participants will be asked to eat soft food and stop tooth brushing (Ezzeldin et al., 2024).
  Arms: 5% NaF fluoride varnish
Other: PRG Barrier coat — Before the application of the varnish, teeth were cleaned using a prophylaxis polishing past with a low-speed cone brush in a contra angle low-speed handpiece. It was then dried with air and isolated using cotton rolls.
  | P a g e 13 According to the manufacturer's instructions, the application of PRG barrier coat varnish a drop of the active will be mixed with the base using the attached brush. After isolation with cotton rolls, the brush will be used to smear the WSLs with the mix. I will be undisturbed for at least three seconds, then cured for 10 seconds using the visible-light curing unit (Ezzeldin etal.,2024).
  And there will be no post operative instruction to patient after application (light cured resin material).
  Arms: PRG Barrier coat

SUMMARY:
To evaluate the remineralization potential of PRG Barrier Coat versus fluoride varnish in white spot lesions in permanent anterior teeth of children.

DETAILED DESCRIPTION:
Dental caries is a complex disease that is very common among children and is increasing rapidly in low- and middle-income countries. The first sign that the caries process has begun is the appearance of localized areas of enamel demineralization, which manifest as white spot lesions (WSL) with varying degrees of opacity. The approach to managing caries is shifting towards a minimally invasive method, focusing on the prevention, reduction, and reversal of caries in its early stages.

By restoring equilibrium between demineralization and remineralization, WSL can be reversed, unlike cavitated carious lesions. The most effective methods for managing and preventing WSLs are those based on fluoride.

Although fluorides have minimal effect on reducing existing WSL, they do prevent the creation of new WSL. Their impact is limited to the enamel's outermost 50 μm layer and does not encourage remineralization across the demineralized lesion body. Visually, the WSL remains nearly unaltered.

Recently S-PRG filler containing material are available., S-PRG fillers have the ability to release and recharge fluoride , S-PRG fillers releases Al, B, Na, Si and Sr ions Silicate and fluoride strongly induce remineralization of the dentin matrix. Strontium and fluoride also improve the acid resistance of teeth by converting hydroxyapatite to strontium apatite and fluoroapatite. S-PRG fillers become available for use in caries prevention where it is hoped that it would enhance mineralization and reduce acidic attack by oral cariogenic bacteria.

According to they concluded that Varnish containing 40% of S-PRG fillers was more effective than the typical 5% NaF-based product and could be used as a substitute for fluoride for the remineralization of initial enamel caries. According to they concluded that S-PRG Barrier Coat has shown better results for treating white spot lesions after one month interval than 5%NaF.

The unique advantage of PRG product (PRG Barrier Coat, SHOFU) is being light-cured, which serves in facilitating the clinical procedure, offering easier application, and adding excellent self-adhesive properties for durable prolonged protection.

To our knowledge there is limited evidence about the clinical performance of PRG barrier coat versus fluoride varnish on white spot lesions remineralization in permanent anterior teeth of children therefore comes the importance of our clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8-14 years with good health according to the American Society of Anesthesiologists (ASA-I).
* Have at least one white spot lesion with International Caries Detection and Assessment System (ICDAS II) score one or two
* Has not used any remineralizing agent in the former three months.
* Parents who accept to sign informed consent.
* Cooperative patients

Exclusion Criteria:

* Patients have caries or restorations in the labial surface.
* Extrinsic or intrinsic stains.
* patients under active orthodontic treatment.
* Uncooperative patient.
* Parents refuse to sign informed consent.
* Medically unfit (other than ASAI).

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Remineralization potential ΔE: will be recorded by the differences in color perception by Spectrophotometer | 1-3-6 months
  The name of measurement: CIELAB parameters, which will record the difference in color perception.
  The CIELAB, or CIE L* a* b*, color system represents quantitative relationship of colors on three axes.
  The measurement tool: spectrophotometer. (L*a*b* values) L*: denoted the tooth lightness.
  1. : indicated hues change across the red-green axis.
  2. : represents hues difference across the yellow-blue axis.

SECONDARY OUTCOMES:
ΔE 2000 will be recorded by Spectrophotometer | 1-3-6 months
  ΔE 2000 will evaluate color difference.
  kL, kC, and kH are parametric coefficients that allow users to adjust the weighting of lightness, chroma, and hue differences, respectively.
  kL: This coefficient controls the weighting of the lightness difference (ΔL*) component in the color difference calculation.
  kC: This coefficient controls the weighting of the chroma difference (ΔC*) component.
  kH: This coefficient controls the weighting of the hue difference (ΔH*) component.

CONTACTS AND LOCATIONS:
Overall Officials: Hala M. Abbas, PhD, Study Director — Head of Department of Pediatric Dentistry and Dental Public Health, Faculty of Dentistry, Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ezzeldin, N., Wahied, D. M., Atef, R., & Mustafa, S. (2024). Clinical evaluation of PRG Barrier coat versus fluoride varnish on the color improvement of white spot lesions in permanent teeth of children: A randomized controlled trial. MSA Dental Journal. https://msadj.journals.ekb.eg/
- [Background] Arifa MK, Ephraim R, Rajamani T. Recent Advances in Dental Hard Tissue Remineralization: A Review of Literature. Int J Clin Pediatr Dent. 2019 Mar-Apr;12(2):139-144. doi: 10.5005/jp-journals-10005-1603. PMID 31571787
- [Background] Amaechi BT, van Loveren C. Fluorides and non-fluoride remineralization systems. Monogr Oral Sci. 2013;23:15-26. doi: 10.1159/000350458. Epub 2013 Jun 28. PMID 23817057
- [Background] Okamoto M, Ali M, Komichi S, Watanabe M, Huang H, Ito Y, Miura J, Hirose Y, Mizuhira M, Takahashi Y, Okuzaki D, Kawabata S, Imazato S, Hayashi M. Surface Pre-Reacted Glass Filler Contributes to Tertiary Dentin Formation through a Mechanism Different Than That of Hydraulic Calcium-Silicate Cement. J Clin Med. 2019 Sep 11;8(9):1440. doi: 10.3390/jcm8091440. PMID 31514356